CLINICAL TRIAL: NCT04009122
Title: Evaluation of the Quality of Life of Patients With Metastatic Non-small Cell Lung Cancer With Supplementary Therapy With IGEN-0206
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igen BioLab SLU (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGEN0206-15
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life of Patients; Non-small Cell Lung Cancer Metastatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IGEN-0206 (Experimental): a sachet after each meal, preferably (3 sachets per day)
  Interventions: Dietary Supplement: IGEN0206
- Placebo (Placebo Comparator): a sachet after each meal, preferably (3 sachets per day)
  Interventions: Other: Placebo
- group C (No Intervention): standard treatment

INTERVENTIONS:
Dietary Supplement: IGEN0206 — Group A
  Arms: IGEN-0206
Other: Placebo — Group B
  Arms: Placebo

SUMMARY:
A national, multicenter, blind, randomized study of three groups, designed to evaluate the impact on the quality of life of IGEN-0206 (IGEN-0206 is a nutritional product, a food) with nutritional support + standard treatment versus nutritional support + standard treatment versus standard treatment in patients with non-lung cancer metastatic microcytic.

The standard treatment can include any line of active treatment (chemotherapy, immunotherapy, biological therapies or targeted therapies), radiotherapy or nonspecific symptomatic treatment.

It will include 280 patients older than 18 years, who have a life expectancy of less than 9 months, who will receive or not active treatment.

After signing the informed consent and confirmation that the subject meets the eligibility criteria, those will be randomized (2: 2: 1 ratio) to receive treatment:

* Group A (112 patients): patients will receive their standard treatment + nutritional support + IGEN-0206
* Group B (112 patients): patients will receive their standard treatment + nutritional support + placebo.
* Group C (56 patients): patients will receive standard treatment. The allocation will be random 2: 2: 1 and will be stratified according to ECOG 1 versus 2-3, type of oncological treatment (chemotherapy, immunotherapy and / or radiotherapy versus targeted therapies versus symptomatic treatment) and type of cancer (squamous versus not flaky).

The present study seeks to demonstrate that IGEN-0206 improves the quality of life and the nutritional status of patients with non-small cell lung cancer. If an improvement in the quality of life is achieved, this could impact on a reduction in the number of treatment delays / omissions, which could secondarily impact on a response and survival benefit (by improving the relative intensity of the active oncological treatment).

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given informed consent in writing, stating that he / she understands the purpose of the study and the procedures it entails, and that he / she agrees to participate.
* Patient with metastatic non-small cell lung carcinoma confirmed by Pathology.
* Expected life expectancy exceeding 12 weeks.
* Age ≥18 years.
* Functional status of the ECOG 1-3.
* Patients who can consume at least 500 ml per day of the nutritional supplement, added to their diet.
* Patients who do not meet criteria for renal failure: the glomerular filtrate, calculated by local formula, must be ≥60 ml / min / 1.73m2.
* Patients who are willing to communicate the use of nutritional supplements, including oral supplements, vitamins and mineral supplements and / or any food supplement
* Patients who are willing to comply with the protocol procedures after having been thoroughly informed about the treatment, the procedures, reviewing the study methodology and signing the informed consent.
* They speak fluent Spanish in order to be able to complete the questionnaires of the study.
* Potentially fertile women must be negative in a serum pregnancy test performed within 7 days prior to entry into the study. Potentially fertile patients participating in this study should use effective contraceptive methods (eg, abstinence, intrauterine device, oral or injectable contraceptives, double-barrier method, or surgical sterilization) to prevent pregnancy, which they will begin to use as of signature of the informed consent document and whose use will continue until at least 13 weeks after the last dose of the study medication has been administered.

Exclusion Criteria:

* Women who are pregnant and / or breast-feeding.
* Persistence of the toxicity of a previous treatment (grade> 1 of the NCI-CTCAE v. 4.03); However, alopecia and sensory neuropathy of grade ≤ 2 are acceptable, as well as other side effects that do not endanger patient safety in the opinion of the researcher.
* Evidence of severe or uncontrolled systemic disease or concomitant process that, in the opinion of the investigator, makes the participation of the subject in the study inadvisable or compromises compliance with the protocol.
* Dementia or mental state significantly altered that could interfere in the understanding and granting of informed consent.
* Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Impact of IGEN-0206 on quality of life in patients with metastatic lung cancer according to the EORTC QLQ-C30. | 52 weeks
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional
Impact of IGEN-0206 on quality of life in patients with metastatic lung cancer according to the EORTC QLQ-L13 | 52 weeks
  The QLQ-LC13 incorporates one multi-item scale to assess dyspnoea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and haemoptysis.
  All of the scales and single-item measures range in score from 0 to 100. A high score for the scales and single items represents a high level of symptomatology or problems

SECONDARY OUTCOMES:
BMI | 52 weeks
  Compare clinical benefits in terms of body mass index (BMI) in the three treatment arms.
Changes in the microbiota | 12 weeks
  Compare changes in the microbiota profile in terms of microbiota metabolism (faecal samples) in the three treatment arms with proteomics and genomics methods.
Interleukin levels | 52 weeks
  To evaluate the changes in the inflammatory and immune response and to identify immunological biomarkers in the blood with predictive power and prognosis.
Cytokines levels | 52 weeks
  To evaluate the changes in the inflammatory and immune response and to identify immunological biomarkers in the blood with predictive power and prognosis.

OTHER OUTCOMES:
Number of Adverse events | 52 weeks
  To compare adverse events (AEs) in the three treatment groups according to the Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.1.
Progression-free survival | 52 weeks
  Time from randomization until the progression of the disease or death from any cause is documented. To compare the efficacy in terms of response and survival among the three arms of the study.
Overall survival | 52 weeks
  Time elapsed from randomization until death is documented for any reason
Objective response rate | 52 weeks
  The sum of the complete and partial answers
Disease control | 52 weeks
  The sum of stable disease and partial / total response.
Number of oncological treatment interruptions | 52 weeks
  To assess tolerability in terms of interruptions or delays in active oncological treatment by adding IGEN-0206

CONTACTS AND LOCATIONS:
Locations (25):
- Spain (25):
  - Hospital Público Virgen de los Lirios, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complexo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital del Henares, Coslada, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Hospital Universitario Son Llatzer, Palma de Mallorca, Palma
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario San Juan De Alicante, Alicante
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Lucus Augusti, Lugo
  - GenesisCare Madrid, Hospital La Milagrosa, Madrid
  - Hospital Sanitas La Zarzuela, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Severo Ochoa, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided
All collected IPD

REFERENCES:
- [Background] Barber MD. Cancer cachexia and its treatment with fish-oil-enriched nutritional supplementation. Nutrition. 2001 Sep;17(9):751-5. doi: 10.1016/s0899-9007(01)00631-1. PMID 11527672
- [Background] Bunn PA Jr, Kelly K. New chemotherapeutic agents prolong survival and improve quality of life in non-small cell lung cancer: a review of the literature and future directions. Clin Cancer Res. 1998 May;4(5):1087-100. PMID 9607565
- [Background] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771